CLINICAL TRIAL: NCT02852642
Title: Structure and Musculoskeletal Function, Functional Capacity and Quality of Life of Elderly Women in Response to a Plyometric Training Model Based on the Stretch-shortening Cycle
Brief Title: Plyometric Training for Elderly Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, João Pedro Pinho, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PlyoElderly
Record Dates: First submitted 2016-07-22; First posted 2016-08-02 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Healthy
Keywords: power training; plyometric training; functional capacity
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise (Experimental): Power training model based in the potentiation of the stretch-shortening cycle.
  Interventions: Other: Exercise
- Control (No Intervention): Maintaining daily activities

INTERVENTIONS:
Other: Exercise — Plyometric training
  Arms: Exercise

SUMMARY:
Introduction: the physiological aging process induces several structural changes in the musculoskeletal system. These, in turn, result in functional changes that are reflected in the senescent dependency, determining the reduction in their quality of life. Power training has been identified as ideal to mitigate the effects of aging. However, there are indications that an intervention based on the potentiation of the stretch-shortening cycle action is a better choice.

DETAILED DESCRIPTION:
Study hypotheses: the participants of the proposed intervention will increase their bone mineral density, muscle volume, functional capacity and will show some improvement in their gait, as well as in their quality of life. Purposes: the main objective of this study was to propose a training model based in the potentiation of the stretch-shortening cycle action and assess its effects on selected parameters of musculoskeletal morphology, functional capacity and quality of life of elderly women.

ELIGIBILITY:
Inclusion Criteria:

* sedentary women, not using bone alteration medication physically able

Exclusion Criteria:

* attending less than 80% of the intervention sessions and not attending the final evaluation

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Bone microstructure | through study completion, an average of 6 months
  Tibia and radius trabecular and cortical bone density
body composition | through study completion, an average of 6 months
  Lean and fat body mass
gait kinematics | through study completion, an average of 6 months
  toe clearance: minimum vertical distance of the forefoot and the ground during swing phase
balance | through study completion, an average of 6 months
  Center of pressure displacement
function capacity assessment | through study completion, an average of 6 months
  timed up and go test
electromyography gait analysis | through study completion, an average of 6 months
  Knee extensors and flexors muscles co-contraction during the gait cycle

CONTACTS AND LOCATIONS:
Overall Officials: Alberto C Amadio, PhD, Study Director — University of Sao Paulo

IPD SHARING:
Plan to Share IPD: No